CLINICAL TRIAL: NCT04878848
Title: Effectiveness of Proprioceptive Neuromuscular Facilitation Techniques in Patients With Adhesive Capsulitis
Brief Title: Proprioceptive Neuromuscular Facilitation Techniques in Patients With Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Meltem Melda Taşkın, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/04
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Adhesive Capsulitis; Shoulder Pain; Shoulder Frozen
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Within the scope of the research, it is planned to apply a traditional rehabilitation program consisting of stretching and strengthening exercises prepared in accordance with the guidelines for one group, and PNF approaches for the upper extremity and scapula in the other group.
Who Masked: Participant
Masking Description: Evaluations will be made by a single investigator and participants will be blinded to what treatment is being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation Group (Experimental): Participants in the proprioceptive neuromuscular facilitation group will be given a treatment protocol consisting of rhythmic initiation, repeated stretch and hold-relax PNF techniques for upper extremity "flexion-abduction-external rotation" pattern and the scapular patterns of anterior elevation, posterior depression, anterior depression, posterior elevation for a total of 4 weeks, 3 days a week for 45 minutes. Assessments will be applied in the baseline and at the end of 4 weeks.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation Exercises
- Conventional Rehabilitation Group (Experimental): Participants in the conventional rehabilitation group will be given a treatment protocol consisting of stretching, strengthening exercises and joint mobilization techniques for a total of 4 weeks, 3 days a week for 45 minutes. Assessments will be applied in the baseline and at the end of 4 weeks.
  Interventions: Other: Conventional Rehabilitation Group

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation Exercises — Within the scope of proprioceptive neuromuscular facilitation exercises, rhythmic initiation, repeated stretch and hold-relax techniques in the upper extremity flexion-abduction-external rotation pattern and scapular patterns of anterior elevation, posterior depression, anterior depression and posterior elevation will be applied to the participants. In addition to these exercises, functional activities in the flexion-abduction-external rotation pattern such as hair combing, turning over from side lying, wearing a jacket, reaching on the shelf will be performed.
  Arms: Proprioceptive Neuromuscular Facilitation Group
Other: Conventional Rehabilitation Group — Active assisted / active range of motion exercises and Wand exercises will be applied to the participants in the conventional rehabilitation group for flexion, abduction and external rotation movements. Exercises will be applied as 5 repetitions in the first 2 weeks and 10 repetitions in the last 2 weeks. Strengthening exercises will be performed with an elastic band and free weights. Strengthening exercises will be started as 2 sets of 5 repetitions and at the end of the second week, it will be applied as 2 sets of 10 repetitions. In addition to these exercises, glenohumeral distraction, glenohumeral posterior and caudal glide will be applied for joint mobilization and it will show progression at the end of the second week.
  Arms: Conventional Rehabilitation Group

SUMMARY:
Adhesive capsulitis is a condition that causes limitation of function and movement in the shoulder joint and affects many activities of daily life. The clinical indicators of adhesive capsulitis; shoulder pain and progressive global stiffness of the glenohumeral joint, night pains and accompanying sleep disturbances, joint capsule contracture, decrease in synovial fluid, abnormal changes in scapular position, functional limitation and consequently decreased quality of life. When we look at the literature, it is seen that traditional rehabilitation practices aim to improve range of motion and reduce pain caused by capsular contracture. In this context, classical therapeutic exercises consisting of stretching and strengthening, joint mobilization methods, proprioceptive neuromuscular facilitation methods are applied. However, there are limited number of studies investigating the effects of PNF techniques on pain, function and activity limitation. Therefore, within the scope of the research, it is planned to apply a traditional rehabilitation program prepared in accordance with the guidelines for one group, and PNF approaches for the upper extremity and scapula in the other group. Thus, it is aimed to examine the effects of the use of upper extremity and scapula PNF techniques on pain, function, range of motion, proprioception, quality of life, sleep and patient satisfaction compared to traditional exercises in adhesive capsulitis rehabilitation. Exercises will be applied 3 days a week for 4 weeks. Each training session will last 45 minutes. Pain, function, range of motion, proprioception, quality of life and sleep quality evaluations will be performed at the beginning of the study and at the end of 4 weeks.

DETAILED DESCRIPTION:
Adhesive capsulitis is a shoulder pathology characterized by contracture of the glenohumeral joint capsule and progressive pain with loss of range of motion. The disease picture is generally examined in 3 phases as painful phase, freezing phase and thaw phase. It is generally characterized by pain, decreased range of motion, function, activity limitations, night pain and sleep disturbances. Sleep disturbances associated with function, activity limitations and night pain negatively affect the patients' quality of life. In the literature, the success rate of conservative treatment is shown as 90%.

Conservative treatment consists of nonsteroidal anti-inflammatory drugs, corticosteroids, and therapeutic exercises. The purpose of therapeutic exercises in general; to reduce pain, increase range of motion, decrease activity limitations, increase scapulohumeral rhythm by correcting impaired shoulder joint biomechanics and improve function. Proprioceptive neuromuscular facilitation (PNF) is an exercise concept that uses proprioceptors to increase responses of the neuromuscular mechanism, range of motion and muscle activation. PNF techniques are applied to improve muscle strength, endurance, mobility, stability, coordination and neuromuscular control and can be easily adapted to daily life activities.

In the literature, it is aimed to increase the glenohumeral joint movements and regulate the scapulothoracic rhythm in the rehabilitation of adhesive capsulitis. However, the number of studies in the literature comparing upper extremity and scapular PNF patterns with classical exercises targeting the glenohumeral and scapulothoracic joints is limited. For this reason, the aim of the study is to focus on the structures involved in shoulder movements in adhesive capsulitis rehabilitation as a whole, and to examine the effects of the use of upper extremity and scapula PNF techniques on pain, function, range of motion, proprioception, quality of life, sleep and patient satisfaction compared to traditional exercises in patients with a diagnosis of adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with unilateral adhesive capsulitis (stage II-III)
* Being between at the ages of 35-65
* Complaints ongoing for at least 3 months

Exclusion Criteria:

* Rheumatological diseases such as rheumatoid arthritis, ankylosing spondylitis
* Being diagnosed with glenohumeral joint osteoarthritis, rotator cuff injury, radiculopathy
* Neurological diseases such as cerebrovascular accident, multiple sclerosis, Parkinson's disease, thoracic outlet syndrome
* Dislocation, subluxation, fracture, infection, tumor
* History of shoulder surgery
* People who cannot cooperate with physiotherapist and exercises.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-08-03 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand Questionnaire | Baseline and end of weeks 4.
  The Disabilities of the Arm, Shoulder and Hand Questionnaire was developed to measure physical disability and symptoms of the upper extremities in people with upper extremity disorders (hand, wrist, elbow, and shoulder). It is a 30-item scale that addresses difficulty in performing various physical activities that require upper extremity function (physical function, 21 items); symptoms of pain, activity-related pain, tingling, weakness, and stiffness (pain symptoms, 5 items); or impact of disability and symptoms on social activities, work, sleep, and psychological well-being (emotional and social function, 4 items). The score ranges from 0 to 100, where 0 = no disability and 100 = most severe disability. In this study, the change that occurred during the 4-week period from the beginning will be examined.

SECONDARY OUTCOMES:
Evaluation of Shoulder Proprioception with Cybex Humac Norm II Isokinetic Dynamometer | Baseline and end of weeks 4.
  Evaluation of shoulder proprioception will be made with Cybex isokinetic device. Measurements will be performed in 30, 60, 90º flexion and abduction and 15, 30º external rotation. For each measurement, the device will be operated 3 times in continuous passive movement (CPM) mode with an angular velocity of 60˚ / second. The patient will be asked to focus on the movement and remember the angle. The difference between the target angle and the angle reached by the patient will be recorded. In this study, the change that occurred during the 4-week period from the beginning will be examined.
Visual Analog Scale | Baseline and end of weeks 4.
  The Visual Analog Scale is a self-reported scale consisting of a horizontal or vertical line, usually 10 centimetres long (100 mm) anchored at the extremes by two verbal descriptors referring to the pain status. The Visual Analogue Scale is a scale in which the severity of pain is marked on a vertical or horizontal line of 0-10 cm in length. During the evaluation, in the measurement of pain intensity, "0: no pain" and "10: unbearable pain" will be explained to the patient. Patients will be asked to mark the level of pain they feel at rest, during activity and at night. In this study, the change that occurred during the 4-week period from the beginning will be examined.
Shoulder Pain and Disability Index | Baseline and end of weeks 4.
  Shoulder, Pain and Disability Index were used to evaluate the functional status of the patients. SPADI is a scale that evaluates the pain and difficulty experienced by patients during various activities. It has 2 different subscales, pain and disability. In the pain subscale, pain status is questioned during 5 different daily life activities. In the disability subscale, the difficulty experienced in 8 different activities is measured. The patient was asked to score the level of pain and difficulty between 0-10 and the values were recorded. (0: no pain, 10: worst imaginable pain - 0: no difficulty, 10: extremely difficult, need help) In this study, the change that occurred during the 4-week period from the beginning will be examined.
Shoulder Disability Scale | Baseline and end of weeks 4.
  Shoulder Disability Scale will be used to assess the disability status associated with pain in the shoulder. The scale includes 16 questions about daily life activities that increase symptoms. Answers to the questions are given as "yes", "no" or "not applicable" depending on whether the activity has been painful in the last 24 hours. The score is calculated by dividing the number of yeses by the sum of the number of yes and the number of no. The obtained score is multiplied by 100 and converted into a percentage value. High score is associated with increased disability. In this study, the change that occurred during the 4-week period from the beginning will be examined.
Range of Motion Assesment | Baseline and end of weeks 4.
  The shoulder flexion, extension, abduction, external and internal rotation openings of the patients will be measured passively and actively with the universal goniometer. Measurements will be made 3 times and the average of each measurement will be recorded. In this study, the change that occurred during the 4-week period from the beginning will be examined.
Lateral Scapular Slide Test | Baseline and end of weeks 4.
  The lateral scapular slide test is a method used for the assessment of dominant and non-dominant side scapular dyskinesia based on the measurement of the distance between the inferior end of the scapula and the spinous process of the vertebra in the same alignment. The difference between the two sides is measured with a tape measure when the arms are at the side of the body and in the resting position, when the hands are at the waist and when the arm is in 90º abduction. Scapular dyskinesia will be considered positive for cases where the distance between the two sides is 1.5 cm or more. In this study, the change that occurred during the 4-week period from the beginning will be examined.
Pittsburgh Sleep Quality Index | Baseline and end of weeks 4.
  Pittsburgh Sleep Quality Index is a self-report scale that determines sleep quality, type and severity of sleep disorder in the last 1 month. Self-report questions include different factors related to sleep quality and these factors are grouped into 7 components. These components are; It provides information on subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills and daytime sleep dysfunction. The total PUKI score takes a value between 0-21. Sleep quality of those with a total score of 5 or less is considered as "healthy", between 6-10 as "bad sleep", and those with a score above 10 as "sleep disorder". In this study, the change that occurred during the 4-week period from the beginning will be examined.
World Health Organization Quality of Life Evaluation Questionnaire Short Form Turkish Version | Baseline and end of weeks 4.
  The health-related quality of life scale was developed by the World Health Organization and aims to evaluate the overall quality of life. The scale consists of 27 questions that measure physical, mental, social and environmental well-being. Since each field expresses the quality of life in its field independently of each other, domain scores are calculated between 4-20. The higher the score means the higher the quality of life. In this study, the change that occurred during the 4-week period from the beginning will be examined.
Global Rating of Change | End of weeks 4.
  It is a widely used scale to evaluate satisfaction in clinical trials, especially in global musculoskeletal problems. It aims to evaluate the effect of treatment and recovery on the patient. The difference between pre-treatment and post-treatment is evaluated on a 5-point numerical scale (-2: much worse, -1: I am worse, 0: I am the same, 1: I am better, 2: I am much better) In this study, we will evaluate patient satisfaction at the end of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yonca Zenginler Yazgan, Assistant Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Demographic informations such as age, gender, height, weight, occupation Results of range of motion, pain severity, function, proprioception, sleep quality, quality of life assessments will be shared with other researches.

REFERENCES:
- [Background] Celik D, Kaya Mutlu E. Does adding mobilization to stretching improve outcomes for people with frozen shoulder? A randomized controlled clinical trial. Clin Rehabil. 2016 Aug;30(8):786-94. doi: 10.1177/0269215515597294. Epub 2015 Jul 30. PMID 26229109
- [Background] Mulligan EP, Brunette M, Shirley Z, Khazzam M. Sleep quality and nocturnal pain in patients with shoulder disorders. J Shoulder Elbow Surg. 2015 Sep;24(9):1452-7. doi: 10.1016/j.jse.2015.02.013. Epub 2015 Apr 1. PMID 25842028
- [Background] Fernandes MR. Correlation between functional disability and quality of life in patients with adhesive capsulitis. Acta Ortop Bras. 2015 Mar-Apr;23(2):81-4. doi: 10.1590/1413-78522015230200791. PMID 27069405
- [Background] Balci NC, Yuruk ZO, Zeybek A, Gulsen M, Tekindal MA. Acute effect of scapular proprioceptive neuromuscular facilitation (PNF) techniques and classic exercises in adhesive capsulitis: a randomized controlled trial. J Phys Ther Sci. 2016 Apr;28(4):1219-27. doi: 10.1589/jpts.28.1219. Epub 2016 Apr 28. PMID 27190456
- [Background] Shimura K, Kasai T. Effects of proprioceptive neuromuscular facilitation on the initiation of voluntary movement and motor evoked potentials in upper limb muscles. Hum Mov Sci. 2002 Apr;21(1):101-13. doi: 10.1016/s0167-9457(01)00057-4. PMID 11983436
- [Background] Toprak M, Erden M. Sleep quality, pain, anxiety, depression and quality of life in patients with frozen shoulder1. J Back Musculoskelet Rehabil. 2019;32(2):287-291. doi: 10.3233/BMR-171010. PMID 30347591
- [Background] Levine WN, Kashyap CP, Bak SF, Ahmad CS, Blaine TA, Bigliani LU. Nonoperative management of idiopathic adhesive capsulitis. J Shoulder Elbow Surg. 2007 Sep-Oct;16(5):569-73. doi: 10.1016/j.jse.2006.12.007. Epub 2007 May 24. PMID 17531513
- [Background] Beaton DE, Katz JN, Fossel AH, Wright JG, Tarasuk V, Bombardier C. Measuring the whole or the parts? Validity, reliability, and responsiveness of the Disabilities of the Arm, Shoulder and Hand outcome measure in different regions of the upper extremity. J Hand Ther. 2001 Apr-Jun;14(2):128-46. PMID 11382253
- [Background] Hayes K, Walton JR, Szomor ZR, Murrell GA. Reliability of five methods for assessing shoulder range of motion. Aust J Physiother. 2001;47(4):289-94. doi: 10.1016/s0004-9514(14)60274-9. PMID 11722295
- [Background] Kibler WB, Sciascia A. Evaluation and Management of Scapular Dyskinesis in Overhead Athletes. Curr Rev Musculoskelet Med. 2019 Dec;12(4):515-526. doi: 10.1007/s12178-019-09591-1. PMID 31760624
- [Background] Ager AL, Roy JS, Roos M, Belley AF, Cools A, Hebert LJ. Shoulder proprioception: How is it measured and is it reliable? A systematic review. J Hand Ther. 2017 Apr-Jun;30(2):221-231. doi: 10.1016/j.jht.2017.05.003. PMID 28641738
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Roach KE, Budiman-Mak E, Songsiridej N, Lertratanakul Y. Development of a shoulder pain and disability index. Arthritis Care Res. 1991 Dec;4(4):143-9. PMID 11188601